CLINICAL TRIAL: NCT05107765
Title: Effects of Pioglitazone on Stress Reactivity and Alcohol Craving
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jin Ho Yoon, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-18-0922 (main study); 1R21AA027273-01A1 (NIH)
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol; Pioglitazone; Stress; Anxiety
MeSH Terms: conditions — Alcoholism; Anxiety Disorders | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pioglitazone (Experimental)
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — For the current trial we will follow recommended adult initial dosing at 30 mg/d to reach maintenance dose of 45 mg/d by end of week 1, which is within standard titration parameters as per the investigator's brochure.
  Arms: Pioglitazone
Drug: Placebo — Pill capsules will look same as that of active drug.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of pioglitazone on stress-induced relapse risk in a laboratory model and to examine the effects of pioglitazone on drinking, stress/anxiety, and alcohol craving in the natural environment

ELIGIBILITY:
Inclusion Criteria:

* treatment-seeking individuals diagnosed with Alcohol Use Disorder Diagnostic (AUD) and Statistical Manual of Mental Disorders, 5th Edition (DSM-5)
* fluent in English
* past month excessive alcohol use (>7 drinks/week for woman, >14 drinks/week for men, >3 drinks/occasion for women>4 drinks/occasion for men)
* exhibit baseline measures of either 1) 8-23 on HAM-A indicative of mild to moderate anxiety, 2) 14-26 on PSS Score indicative of moderate stress, or 3) ≥2 on Drinking Motives Questionnaire (DMQ-R) questions related to drinking indicating that individuals drink at least "some of the time" to cope
* exhibit increased stress reactivity (increased physiological response and/or self-report) at the baseline stress reactivity assessment
* females will need to agree to use of barrier methods of contraception due to pioglitazone's effects on plasma concentrations of oral contraceptives

Exclusion Criteria:

* Exhibit severe scores on the HAM-A, PSS, or PTSD checklist (PCL-5) - may be enrolled at the discretion of the admitting physician (Dr. Weaver)
* physical dependence on alcohol (CIWAA > 10)
* greater than mild substance use disorder on drugs other than alcohol, nicotine, and marijuana
* contraindications for taking pioglitazone
* medical conditions (e.g., congestive heart failure, clinically significant edema, clinically significant liver disease, hypoglycemia, diabetes, history of bladder cancer)
* contraindicating pioglitazone pharmacotherapy or taking contraindicated medications (e.g., CYP2C8 inhibitors or inducers, antihyperglycemic medications)
* be pregnant, nursing, or planning on becoming pregnant during the course of the study
* have any other illness, condition, or use of medications, which in the opinion of the PI and/or admitting physician would preclude safe and/or successful completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin H Yoon, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 67 participants enrolled, 55 were randomized; 8 were lost to follow-up before randomization, and 4 withdrew before randomization.
Period: Overall Study
Arm/Group | Placebo | Pioglitazone
Started | 29 | 26
Completed | 18 | 22
Not Completed | 11 | 4
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawn by investigator due to non-compliance | 1 | 0
Not completed — Withdrawal by Subjects due to scheduling issues | 6 | 3

BASELINE CHARACTERISTICS:
Population: Includes all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pioglitazone | Total
Number analyzed (Participants) | 29 | 26 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.03 (13.63) | 33.58 (10.26) | 35.93 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 19 | 17 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 17 | 15 | 32
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 29 | 26 | 55
Years of Education [Mean (Standard Deviation); unit: years] | 15.38 (1.92) | 15.92 (2.9) | 15.64 (2.12)

OUTCOME MEASURES:

1. Primary Outcome: Change in Stress-reactivity as Assessed by Heart Rate Change During the Cold Pressor Task (CPT)
Description: During the cold pressor task (CPT), participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. Heart rate will be collected before and after CPT. The change in Heart rate will be reported as [(Heart rate post cold pressor task) - (Heart rate pre cold pressor task)].
Time Frame: Baseline, about 2 minutes after the start of the cold pressor task
Measure: Mean (Standard Deviation); unit: beats per minutes (bpm)
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 29 | 26
beats per minutes (bpm) | 5.138 (11.426) | 12.154 (11.885)

2. Primary Outcome: Change in Stress-reactivity as Assessed by Heart Rate Change During the Cold Pressor Task (CPT)
Description: as for outcome 1
Time Frame: Week 8, about 2 minutes after the start of the Cold Pressor Task
Measure: Mean (Standard Deviation); unit: beats per minutes (bpm)
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 18 | 22
beats per minutes (bpm) | 4.444 (8.118) | 11.182 (12.945)

3. Primary Outcome: Change in Stress-reactivity as Assessed by Change in Systolic Blood Pressure During the Cold Pressor Task (CPT)
Description: During the cold pressor task (CPT), participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. Systolic Blood Pressure will be collected before and after CPT. The change in Systolic Blood Pressure will be reported as [( Systolic Blood Pressure at post cold pressor task) - (Systolic Blood Pressure at pre cold pressor task)].
Time Frame: Baseline, about 2 minutes after the start of the Cold Pressor Task
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 29 | 26
millimeters of mercury (mmHg) | 19.931 (12.236) | 20.038 (13.721)

4. Primary Outcome: Change in Stress-reactivity as Assessed by Change in Systolic Blood Pressure During the Cold Pressor Task (CPT)
Description: as for outcome 3
Time Frame: Week 8, about 2 minutes after the start of the Cold Pressor Task
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 18 | 22
millimeters of mercury (mmHg) | 17.778 (10.963) | 21.091 (15.165)

5. Primary Outcome: Change in Stress-reactivity as Assessed by Diastolic Blood Pressure Change During the Cold Pressor Task (CPT)Cold Pressor Task (CPT)
Description: During the cold pressor task (CPT), participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. Diastolic Blood Pressure will be collected before and after CPT. The change in Diastolic Blood Pressure will be reported as [( Diastolic Blood Pressure post cold pressor task) - (Diastolic Blood Pressure pre cold pressor task)].
Time Frame: Baseline, about 2 minutes after the start of the Cold Pressor Task
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 29 | 26
millimeters of mercury (mmHg) | 12.793 (8.862) | 13.192 (10.257)

6. Primary Outcome: Change in Stress-reactivity as Assessed by Diastolic Blood Pressure Change During the Cold Pressor Task (CPT)Cold Pressor Task (CPT)
Description: as for outcome 5
Time Frame: Week 8, about 2 minutes after the start of the Cold Pressor Task
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 18 | 22
millimeters of mercury (mmHg) | 12 (9.911) | 13.545 (10.613)

7. Primary Outcome: Change in Stress-reactivity as Assessed by Salivary Cortisol Level Change During the Cold Pressor Task (CPT)
Description: During the cold pressor task (CPT), participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. Saliva samples will be collected before and after the CPT, and cortisol levels in the saliva samples will be assessed. The change in cortisol level will be reported as [(cortisol level at post cold pressor task) - (cortisol level pre cold pressor task)].
Time Frame: baseline, about 32 minutes after the start of the Cold Pressor Task
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 29 | 26
picograms per milliliter (pg/mL) | 230.087 (1040.858) | 908.96 (2046.185)

8. Primary Outcome: Change in Stress-reactivity as Assessed by Salivary Cortisol Level Change During the Cold Pressor Task (CPT)
Description: as for outcome 7
Time Frame: week 8, about 32 minutes after the start of the Cold Pressor Task
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 18 | 22
picograms per milliliter (pg/mL) | 427.61 (917.927) | 447.417 (1466.214)

9. Primary Outcome: Change in Alcohol Craving as Assessed by Alcohol Craving Scale Score During the Cold Pressor Task (CPT)
Description: The alcohol craving scale has a total score from 0 to 50, higher score indicating greater alcohol craving. During the cold pressor task (CPT), participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. The Alcohol Craving Scale will be administered before and after CPT. The change in alcohol craving will be reported as [(Alcohol craving scale score post cold pressor task) - (Alcohol craving scale score pre cold pressor task)]. -- a negative value indicates a decrease in alcohol craving.
Time Frame: baseline, about 2 minutes after the start of the CPT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 29 | 26
score on a scale | -0.083 (1.36) | 0.092 (1.877)

10. Secondary Outcome: Change in Drinking Habit as Assessed by the Number of Drinks Per Day (Timeline Followback Method)
Description: The Timeline Followback (TLFB) method was used to assess alcohol consumption by asking study participants to self-report their number of drinks consumed each day over the past week.
  The change in drinking habit is reported as [(number of drinks per day at week 8) - (number of drinks per day at baseline)].-- a negative value indicates a decrease in alcohol consumption over time.
Time Frame: baseline, week 8
Measure: Mean (Standard Deviation); unit: drinks per day
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 18 | 22
drinks per day | -1.229 (1.49) | -0.714 (1.02)

11. Secondary Outcome: Change in Drinking Habit as Assessed by the Number of Heavy Drinking Days (Timeline Followback Method)
Description: The Timeline Followback (TLFB) method was used to assess alcohol consumption by asking study participants to self-report their number of drinks consumed each day over the past week.
  Heavy drinking is defined as 4 drinks or more per day for females and 5 or more drinks per day for males. The change in drinking habit is reported as [(number of heavy drinking days at week 8) - (number of heavy drinking days at baseline)].--A negative value indicates a decrease in the number of heavy drinking days over time.
Time Frame: baseline, week 8
Measure: Mean (Standard Deviation); unit: Heavy drinking days
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 18 | 22
Heavy drinking days | -5.5 (5.113) | -3.591 (4.152)

12. Secondary Outcome: Anxiety as Assessed by the Hamilton Anxiety Rating Scale(HAM-A)
Description: The Hamilton Anxiety Rating Scale(HAM-A) is a 14 item questionnaire scored from 0 (not present) to 4 (very severe). The 14 items are summed to obtain a total score ranging from 0 to 56, high scores indicating greater anxiety.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 29 | 26
score on a scale | 5.862 (4.991) | 4 (3.929)

13. Secondary Outcome: Anxiety as Assessed by the Hamilton Anxiety Rating Scale(HAM-A)
Description: as for outcome 12
Time Frame: week 1
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 24 | 24
score on a scale | 5.458 (5.141) | 3.458 (3.538)

14. Secondary Outcome: Anxiety as Assessed by the Hamilton Anxiety Rating Scale(HAM-A)
Description: as for outcome 12
Time Frame: week 2
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 23 | 23
score on a scale | 4.087 (4.01) | 3.435 (3.116)

15. Secondary Outcome: Anxiety as Assessed by the Hamilton Anxiety Rating Scale(HAM-A)
Description: as for outcome 12
Time Frame: week 3
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 22 | 21
score on a scale | 4.727 (4.143) | 2.95 (3.236)

16. Secondary Outcome: Anxiety as Assessed by the Hamilton Anxiety Rating Scale(HAM-A)
Description: as for outcome 12
Time Frame: week 4
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 20 | 21
score on a scale | 4.1 (4.291) | 2.524 (4.308)

17. Secondary Outcome: Anxiety as Assessed by the Hamilton Anxiety Rating Scale(HAM-A)
Description: as for outcome 12
Time Frame: week 5
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 20 | 22
score on a scale | 3.45 (4.019) | 2.5 (2.502)

18. Secondary Outcome: Anxiety as Assessed by the Hamilton Anxiety Rating Scale(HAM-A)
Description: as for outcome 12
Time Frame: week 6
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 20 | 21
score on a scale | 2.895 (3.053) | 2.6 (3.662)

19. Secondary Outcome: Anxiety as Assessed by the Hamilton Anxiety Rating Scale(HAM-A)
Description: as for outcome 12
Time Frame: week 7
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 20 | 22
score on a scale | 2.842 (2.566) | 3.364 (5.876)

20. Secondary Outcome: Anxiety as Assessed by the Hamilton Anxiety Rating Scale(HAM-A)
Description: as for outcome 12
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 18 | 22
score on a scale | 4.167 (3.869) | 2.952 (4.226)

21. Secondary Outcome: Alcohol Craving as Assessed by the Pennsylvania Alcohol Craving Scale(PACS)
Description: The Pennsylvania Alcohol Craving Scale(PACS) total score ranges from 0 to 30, higher scores indicating more alcohol cravings.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 29 | 26
score on a scale | 11.103 (4.678) | 9.577 (5.994)

22. Secondary Outcome: Alcohol Craving as Assessed by the Pennsylvania Alcohol Craving Scale(PACS)
Description: as for outcome 21
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 18 | 22
score on a scale | 5.6111 (5.6375) | 7.409 (5.981)

23. Secondary Outcome: Stress as Assessed by the Perceived Stress Scale(PSS)
Description: The Perceived Stress Scale(PSS) is a 10 item questionnaire scored from 0 (never) to 4 (very often). The 10 items are summed to obtain a total score ranging from 0 to 40, high scores indicating greater stress.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 29 | 26
score on a scale | 14.276 (7.892) | 12.808 (7.731)

24. Secondary Outcome: Stress as Assessed by the Perceived Stress Scale(PSS)
Description: as for outcome 23
Time Frame: Week 1
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 24 | 24
score on a scale | 15.208 (7.407) | 14.583 (6.928)

25. Secondary Outcome: Stress as Assessed by the Perceived Stress Scale(PSS)
Description: as for outcome 23
Time Frame: Week 2
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 23 | 23
score on a scale | 13.522 (7.988) | 14.783 (6.915)

26. Secondary Outcome: Stress as Assessed by the Perceived Stress Scale(PSS)
Description: as for outcome 23
Time Frame: Week 3
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 22 | 21
score on a scale | 13.318 (6.785) | 14.19 (8.116)

27. Secondary Outcome: Stress as Assessed by the Perceived Stress Scale(PSS)
Description: as for outcome 23
Time Frame: Week 4
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 20 | 21
score on a scale | 12.65 (9.08) | 14.143 (6.24)

28. Secondary Outcome: Stress as Assessed by the Perceived Stress Scale(PSS)
Description: as for outcome 23
Time Frame: Week 5
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 20 | 22
score on a scale | 12.55 (8.787) | 12.227 (7.237)

29. Secondary Outcome: Stress as Assessed by the Perceived Stress Scale(PSS)
Description: as for outcome 23
Time Frame: Week 6
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 20 | 21
score on a scale | 13.8 (6.478) | 12.429 (7.427)

30. Secondary Outcome: Stress as Assessed by the Perceived Stress Scale(PSS)
Description: as for outcome 23
Time Frame: Week 7
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 20 | 22
score on a scale | 11.7 (5.966) | 12.455 (8.629)

31. Secondary Outcome: Stress as Assessed by the Perceived Stress Scale(PSS)
Description: as for outcome 23
Time Frame: Week 8
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 18 | 22
score on a scale | 11.222 (7.224) | 12.318 (6.284)

32. Primary Outcome: Change in Alcohol Craving as Assessed by Alcohol Craving Scale Score During the Cold Pressor Task (CPT)
Description: as for outcome 9
Time Frame: week 8, about 2 minutes after the start of the CPT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 18 | 22
score on a scale | 0.367 (0.963) | 1.173 (2.196)

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Arm/Group | Placebo | Pioglitazone
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/26
Other Adverse Events (participants affected / at risk) | 25/29 | 22/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | Pioglitazone (N=26)
Drowsiness (Nervous system disorders) | 12 | 11
Not Sleeping Well (Nervous system disorders) | 13 | 12
Headache (Nervous system disorders) | 8 | 11
Nervousness (Nervous system disorders) | 2 | 2
Blurry Vision (Nervous system disorders) | 5 | 1
Dizziness (Nervous system disorders) | 4 | 3
Tremor (Nervous system disorders) | 7 | 7
Sweating (Nervous system disorders) | 6 | 3
Confusion (Nervous system disorders) | 2 | 3
Cloudiness (Nervous system disorders) | 3 | 6
Memory Loss (Nervous system disorders) | 4 | 6
Fatigue Tiredness (Nervous system disorders) | 1 | 0
Difficulty Walking (Nervous system disorders) | 1 | 4
Weakness (Nervous system disorders) | 5 | 5
Heart Racing (Nervous system disorders) | 3 | 3
Chest pain (Nervous system disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 6 | 4
Vomiting (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 6 | 9
Diarrhea (Gastrointestinal disorders) | 3 | 8
Stomach Cramps (Gastrointestinal disorders) | 9 | 7
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Increased Urination (Renal and urinary disorders) | 5 | 4
Dry Mouth (Endocrine disorders) | 10 | 14
Loss of appetite (Endocrine disorders) | 1 | 2
Fever or Chills (Immune system disorders) | 3 | 5
skin rash (Immune system disorders) | 4 | 3
Muscle Aches (Musculoskeletal and connective tissue disorders) | 5 | 5
Elevated CK Levels (Musculoskeletal and connective tissue disorders) | 2 | 0
Swelling (Blood and lymphatic system disorders) | 1 | 3
Change in Sexual Function (Reproductive system and breast disorders) | 5 | 3

LIMITATIONS AND CAVEATS:
Due to technical problems, the data for the outcome measure "Change in Stress-reactivity as Assessed by Salivary Cortisol Level Change During the Cold Pressor Task (CPT)" at both baseline and Week 8 were found to be unreliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT05107765/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT05107765/ICF_001.pdf